CLINICAL TRIAL: NCT04987255
Title: The Art of Moving for Sustainable Health: Influence of a Museum Visit on the Physical Demands and Well-being of Sedentary People
Brief Title: The Art of Moving for Sustainable Health
Acronym: ART-M2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: School of Health Sciences Geneva (Other)
Responsible Party: Principal Investigator, Anne-Violette Bruynnel, Professor, School of Health Sciences Geneva
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 112187
Record Dates: First submitted 2021-07-21; First posted 2021-08-03 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Sedentary Behavior; Stroke
Keywords: Physical activity; Museum; Well-being; Sedentary; Stroke
MeSH Terms: conditions — Sedentary Behavior; Stroke; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Free visit (Active Comparator): Free visit of the museum during 75 minutes for individuals in sedentary condition (healthy)
  Interventions: Other: Free visit
- Guided visit (Experimental): Guided visit of the museum during 75 minutes for individuals in sedentary condition (healthy)
  Interventions: Other: Guided visit
- Guided visit for individuals after stroke (Other): This arm is specific for individuals with motor disability after stroke (non randomized condition)
  Interventions: Other: Guided visit (stroke)

INTERVENTIONS:
Other: Free visit — The persons with sedentary (healthy) in this group will have to visit the museum freely (without a guide) for a period of 75 minutes.
  Arms: Free visit
Other: Guided visit — The persons with sedentary (healthy) in this group will have to visit the museum with a guide for a period of 75 minutes.
  Arms: Guided visit
Other: Guided visit (stroke) — The persons with motor disability after stroke in this group will have to visit the museum with a guide for a period of 75 minutes.
  Arms: Guided visit for individuals after stroke

SUMMARY:
Sedentary behaviour is particularly high among the older and in the presence of a chronic pathology. Physical activity is limited mainly by the lack of accessibility to activities offered in the city and the lack of motivation.

The objective is to study the physical solicitations and the well-being during the visit of a museum (free or guided visit). Our hypothesis is that this cultural activity induces a sufficient physical solicitation for sedentary people and for individuals with a post-stroke motor disability.

All the tests will be carried out during the same day by experienced physiotherapists. Physical and well-being tests will be performed before and after the visits. The number of steps taken during the visit will be measured.

This is a different approach to promote physical activity and this proposal is an original way to stimulate the physical, psychic and social health of sedentary people. If the results are beneficial, museums could become real health partners to stimulate the activity of sedentary people.

ELIGIBILITY:
Inclusion Criteria:

* Age > 50 years
* Sedentary condition (<150 minutes of physical activity per week)
* Medical stability
* Mini Mental State Evauation > 22
* Walking independently with or without assistance
* MiniBESTest > 20/28
* For individuals with stroke: chronic post-stroke condition.

Exclusion Criteria:

* Refusal to participate;
* Person with other conditions affecting independent walking;
* Contraindications to prolonged standing;
* Pain greater than 4/10 on the NRS;
* Concomitant pathologies that may interfere with the results;
* Inability to follow the study procedure (cognitive disorders, dementia, psychological disorders, language problems...).

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2023-03-14 (Actual); Study Completion 2023-03-14 (Actual)

PRIMARY OUTCOMES:
Number of steps during visit in the three groups (free visit vs. guided visit and guided visit for individuals with stroke) | 75 minutes
  An activity tracker on the visitor's wrist will measure the number of steps taken while visiting the museum. Parameter: number of steps.

SECONDARY OUTCOMES:
Change from baseline (pre-visit): Postural control in the three groups (free visit vs. guided visit and guided visit for individuals with stroke) | 75 minutes
  The standing balance will be tested in bipedal with forceplate. Parameters: center of pressure displacement (mm).
Change from baseline (pre-visit): Postural control in the three groups (free visit vs. guided visit and guided visit for individuals with stroke) | 75 minutes
  The standing balance will be tested in bipedal with forceplate. Parameters: center of pressure speed (mm/s).
Change from baseline (pre-visit): Postural control in the three groups (free visit vs. guided visit and guided visit for individuals with stroke) | 75 minutes
  The standing balance will be tested in bipedal with forceplate. Parameters: center of pressure sway area (mm2).
Change from baseline (pre-visit): gait speed in the three groups (free visit vs. guided visit and guided visit for individuals with stroke) | 75 minutes
  The gait speed will be tested with the Ten-meter walking test. Parameter: gait speed (m/s)
Change from baseline (pre-visit): sit to stand transfert in the three groups (free visit vs. guided visit and guided visit for individuals with stroke) | 75 minutes
  The sit to stand transfert will be tested with the five sit to stand test. Parameter: duration to realize five sit-to stand transferts (seconds)
Change from baseline (pre-visit): lower limb muscle strength in the three groups (free visit vs. guided visit and guided visit for individuals with stroke) | 75 minutes
  The knee extensors muscle strength will be measured with an hand-held dynamometer. Parameter: maximal voluntary force in Newton (N).
Change from baseline (pre-visit): fatigue in the three groups (free visit vs. guided visit and guided visit for individuals with stroke) | 75 minutes
  The fatigue will be tested with the Numeric Rating Scale. Parameter: 10-points score.
Change from baseline (pre-visit): pain in the three groups (free visit vs. guided visit and guided visit for individuals with stroke) | 75 minutes
  The pain will be tested with the Numeric Rating Scale. Parameter: 10-points score.
Change from baseline (pre-visit): anxiety in the three groups (free visit vs. guided visit and guided visit for individuals with stroke) | 75 minutes
  The anxiety will be tested with the Numeric Rating Scale. Parameter: 10-points score.
Change from baseline (pre-visit): museum well-being in the three groups (free visit vs. guided visit and guided visit for individuals with stroke) | 75 minutes
  The well-being will be tested with the museum well-being survey.
Safety endpoint 1: fatigue | 3 hours
  The fatigue will be tested with the Numeric Rating Scale. Parameter: 10-points score.
Safety endpoint 2: pain | 3 hours
  The fatigue will be tested with the Numeric Rating Scale. Parameter: 10-points score.
Safety endpoint 3: number of subjects | 3 hours
  The safety endpoint will be tested with the calculation of the number of subjects who completed the visit and the tests.

OTHER OUTCOMES:
Cognitive status in the three groups (free visit vs. guided visit and guided visit for individuals with stroke) | baseline 60 minutes
  The cognitive function will be tested with the Mini Mental State Evaluation. Parameter: score / 28 points.
Motor status in the three groups (free visit vs. guided visit and guided visit for individuals with stroke) | baseline 60 minutes
  The motor function will be tested with the Mini BESTest. Parameter: score in percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Anne-violette Bruyneel, Principal Investigator — School of Health Sciences Geneva
Locations (1):
- Musées de la ville de Genève, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measure will be made available.
Supporting Information: Study Protocol
Time Frame: Data will be available within 6 months of study completion
Access Criteria: At the end of the project the data will be deposited in the Yareta repository developed by the University of Geneva OR in an institutional repository. This choice will ensure that data is archived and shared in accordance with FAIR principles.

REFERENCES:
- [Background] Harvey JA, Chastin SF, Skelton DA. Prevalence of sedentary behavior in older adults: a systematic review. Int J Environ Res Public Health. 2013 Dec 2;10(12):6645-61. doi: 10.3390/ijerph10126645. PMID 24317382
- [Background] Tudor-Locke C, Craig CL, Aoyagi Y, Bell RC, Croteau KA, De Bourdeaudhuij I, Ewald B, Gardner AW, Hatano Y, Lutes LD, Matsudo SM, Ramirez-Marrero FA, Rogers LQ, Rowe DA, Schmidt MD, Tully MA, Blair SN. How many steps/day are enough? For older adults and special populations. Int J Behav Nutr Phys Act. 2011 Jul 28;8:80. doi: 10.1186/1479-5868-8-80. PMID 21798044
- [Background] Mastandrea S, Fagioli S, Biasi V. Art and Psychological Well-Being: Linking the Brain to the Aesthetic Emotion. Front Psychol. 2019 Apr 4;10:739. doi: 10.3389/fpsyg.2019.00739. eCollection 2019. PMID 31019480
- [Background] Camic PM, Chatterjee HJ. Museums and art galleries as partners for public health interventions. Perspect Public Health. 2013 Jan;133(1):66-71. doi: 10.1177/1757913912468523. PMID 23308010